CLINICAL TRIAL: NCT01448603
Title: An Optional One Year Follow-up Study to Evaluate the Continued Efficacy of ToleroMune Ragweed in Ragweed Allergic Subjects Following Challenge With Ragweed Allergen in an Environmental Exposure Chamber.
Brief Title: ToleroMune Ragweed Follow up Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Cetero Research, San Antonio (Network)
Responsible Party: Sponsor
Other Study IDs: TR002B
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Ragweed Allergy; Rhinoconjunctivitis
Keywords: Ragweed allergy; ToleroMune ragweed; immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Placebo: Subjects previously randomised to placebo in TR002
  Interventions: Biological: Placebo
- ToleroMune Ragweed Regimen 1: Subjects previously randomised to receive ToleroMune Ragweed regimen 1 in study TR002
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed Regimen 2: Subject previously randomised to receive ToleroMune Ragweed regimen 2 in study TR002
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed regimen 3: Subject previously randomised to receive ToleroMune Ragweed regimen 3 in study TR002
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed regimen 4: Subjects previously randomised to receive ToleroMune Ragweed regimen 4 in study TR002
  Interventions: Biological: ToleroMune Ragweed

INTERVENTIONS:
Biological: Placebo — No further medication to be administered in this study. Intervention refers to treatment received in Study TR002.
  Groups: Placebo
Biological: ToleroMune Ragweed — No further medication to be administered in this study. Intervention refers to treatment received in Study TR002.
  Groups: ToleroMune Ragweed Regimen 1; ToleroMune Ragweed Regimen 2; ToleroMune Ragweed regimen 3; ToleroMune Ragweed regimen 4

SUMMARY:
Ragweed is the primary cause of autumn allergies. The ragweed season begins in mid-August. In the third National Health and Nutrition Examination Surveys54.3% of the population had positive test responses to one or more allergens, with the prevalence for short ragweed being 26.2%

The purpose of this observational follow-on study is to further evaluate rhinoconjunctivitis symptoms on exposure to ragweed allergen in the EEC among subjects who completed all dosing visits and the post treatment challenge (PTC) visit in study TR002 approximately one year after the start of treatment.

DETAILED DESCRIPTION:
Subjects who were randomised in study TR002 and who completed all dosing visits and the PTC will be invited to attend the Screening Visit for TR002B. Subjects will attend the EEC for 4 visits on successive days. Following the final EEC visit a follow-up visit will be performed 3-10 days later.

ELIGIBILITY:
Inclusion Criteria

* Previously randomised into study TR002 and completed all treatment visits and the PTC.

Exclusion Criteria

* History of asthma (a diagnosis of asthma in childhood may be allowed).
* Subjects with an FEV1 <70% of predicted.
* Subjects being treated with beta-blockers.
* Developed a significant disease, disorder or inability to communicate, since completing study TR002 which, in the opinion of the Sponsor's medical representative, may either put the subject at risk because of participation in the study, or influence the results of the study, or the subject's ability to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously randomised in study TR002 and completed all dosing visits and the Post Treatment Challenge (PTC).
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | 48-54 weeks after the start of treatment in TR002

SECONDARY OUTCOMES:
Total nasal and non-nasal symptom scores | 48-54 weeks after the start of treatment in TR002
Change in Immunoglobulin A (IgA) | 50-56 weeks after the start of treatment in Tr002
Change in Immunoglobulin E (IgE) | 50-56 weeks after the start of treatment in Tr002
Change in Immunoglobulin G4 (IgG4) | 50-56 weeks after the start of treatment in Tr002
Adverse Events | 50-56 weeks after the start of treatment in TR002

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada